CLINICAL TRIAL: NCT01903642
Title: Study of the Proteome and Cytokines During Inflammatory Syndromes of Different Etiologies.
Acronym: Proteome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: Bonnotte PHRC IR 2008
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Inflammatory Disease

ARMS (1):
- Patients with inflammatory syndrome (Other)
  Interventions: Other: proteomic analysis

INTERVENTIONS:
Other: proteomic analysis

SUMMARY:
The hypotheses of our research are based on the fact that various pathological states, infection, cancer, inflammatory disease, can induce an inflammatory syndrome, through different pathways, even though the clinical presentation can be identical. The identification of biological markers specific to an etiology would therefore allow a faster diagnosis and improve care for patients. We thus took an interest in the three groups of diseases most frequently responsible for an inflammatory syndrome, infections, cancers and auto-immune diseases. To achieve this, various methods will be used.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting an inflammatory syndrome, defined by elevated C-reactive protein (CRP>50mg/L), whose etiology is related to infection, cancer or an inflammatory disease.

* Patients not on treatment (corticoids, immunosuppressive drugs) during the 7 days preceding inclusion
* Age: 18-90 years
* Patients covered by the National Health Insurance Agency
* signed written informed consent form

Exclusion Criteria:

* - Any patient not meeting the inclusion criteria
* Pregnant patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
determination of usual parameters of inflammation | at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France